CLINICAL TRIAL: NCT06606119
Title: The Role of Brain-Bone Marrow-Gut Interaction Following Major Trauma
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202400903; 1R35GM152216-01 (NIH)
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Trauma Injury; Trauma; Critical Illness; Microbiome; Chronic Anemia; Acute Blood Loss Anemia
Keywords: Hematopoietic Stem Progenitor Cells; Bone Marrow Failure; Anemia; Gut Microbiome; Inflammation; Dysregulated Stress Response
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Critical Illness; Bone Marrow Failure Disorders; Anemia; Inflammation | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow, Blood, Feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major Trauma Injury: Severe blunt trauma patients diagnosed with shock with a long bone or pelvic fracture requiring open reduction internal fixation or intramedullary fixation.
  Interventions: Other: Data and tissue collection
- Elective Hip Replacement: Patients undergoing elective hip replacement surgery
  Interventions: Other: Data and tissue collection

INTERVENTIONS:
Other: Data and tissue collection — Collection of bone marrow, blood, feces, medical record data, and patient response surveys.

SUMMARY:
Traumatic injury followed by critical illness provokes pathophysiologic changes in the bone marrow and the gut that contribute to persistent anemia and changes in the microbiome which significantly impact long-term recovery. This project will define the interactions between the stress, chronic inflammation, bone marrow dysfunction, and an altered microbiome which will provide a strong foundation for future clinical interventions to help improve outcomes following severe trauma.

DETAILED DESCRIPTION:
Trauma remains the leading cause of death among people younger than 46 years of age and is the leading cause of years of potential life lost among those younger than 65. With more lives saved, trauma morbidity has increased, which has consequently revealed a lack of understanding of the impact of trauma survivorship on the patients' quality of life and long-term recovery. Severe injury when followed by chronic critical illness leads to persistent anemia, and the use of blood transfusions is associated with a linear increase in infectious complications. These conditions are due to prolonged bone marrow dysfunction associated with an exaggerated catecholamine response, chronic stress, and systemic inflammation. Our laboratory has conducted human research to establish that there are unique bone marrow transcriptomic differences related to inflammation, the innate immune response, and known inhibitors of erythropoiesis following trauma. The laboratory has also discovered that chronic stress after trauma contributes to persistent anemia with impaired iron and erythropoietin function along with the prolonged loss of hematopoietic stem progenitor cells (HSPC) from the bone marrow. Chronic stress after trauma also induces an altered microbiome with decreased alpha and beta diversity and changes in microbial composition leading to a persistent 'pathobiome'. All of these factors influence outcomes. We hypothesize that there is a unifying interaction between stress, inflammation, and the microbiome and this has an overall role in the regulation of HSPC and erythroid progenitor cell fate and function following trauma and critical illness. Therefore, the overarching goal for this study is to build upon this foundation and expand our understanding of HSPC fate and function following trauma, including examining interventions aimed at reducing stress/inflammation and restoring the microbiome, thus, improving long-term outcomes.

ELIGIBILITY:
Severe Trauma Cohort

Inclusion Criteria:

1. All adults (age ≥18).
2. Blunt trauma with an injury severity score > 15 and a long bone or pelvic fracture requiring open reduction internal fixation or intramedullary fixation
3. Blunt trauma patients with shock, defined by either a systolic BP (SBP) <90 mm Hg or base deficit (BD) ≥5 meq or lactate ≥ 2 mmol/L or active red blood cell or whole blood transfusion within 6h or arrival

Exclusion Criteria:

1. Patients not expected to survive greater than 48 hours
2. Prisoners
3. Pregnancy
4. Previous bone marrow transplantation
5. Patients receiving chronic corticosteroids or immunosuppression therapies
6. Patients with End Stage Renal Disease
7. Patients with any pre-existing hematological disease
8. Surgery for repair of injury is greater than seven days after admission to the hospital for trauma
9. Burn injury greater than 20% TBSA

Elective Hip Cohort

Inclusion Criteria

1. All adults (age ≥55).
2. Patient undergoing elective hip repair for non-infectious reasons.
3. Ability to obtain Informed Consent prior to operation.

Exclusion Criteria

1. Patients not expected to survive greater than 48 hours
2. Prisoners
3. Pregnancy
4. Previous bone marrow transplantation
5. Patients receiving chronic corticosteroids or immunosuppression therapies
6. Patients with End Stage Renal Disease
7. Patients with any pre-existing hematological disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Care Trauma ICU - Severe Blunt Trauma Orthopedic Injury Shock Orthopedic Clinic - Elective Hip Replacement
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Link the changes in HSPC and erythroid progenitor cell fate and function with sympathetic stress-induced changes establishing brain-bone marrow communication following trauma. | 3 years
  The impact of the severity and duration of catecholamine secretion on the cellular biology of HSPCs and erythroid progenitor cells requires further detailed evaluation. At each stage of proliferation and differentiation, there is a complex interaction of cytokines, transcription factors, post-translational modification of histones, and miRs. Single-cell RNA-seq technologies using a novel second generation multi-omics technology, CITE-seq, will be used for identification of isolated HSPCs and erythroid progenitor cells. Such single cell sequencing technology is ideal for cell populations with a great deal of heterogeneity and is well-suited for bone marrow analysis. Isolated cells can then be characterized by their transcriptomic and epigenetic changes. We will also evaluate EVM cargo (specific proteins/RNA/miR) from both plasma and bone marrow to determine links to chronic stress exposure.
Determine the connection between changes in the microbiome with sympathetic stress-induced changes establishing gut-brain communication following trauma. | 3 years
  Focusing on the effects of autonomic nervous system on gut function and immune responses, in the setting of sympathetic activation, a serial evaluation of the gut microbiota and their metabolic products (ex. SCFAs: butyrate, propionate, and acetate) will be performed in trauma patients. Correlation of microbial diversity and alterations of the taxonomic composition will be correlated with plasma markers of inflammation and clinical outcomes. Longitudinal study of the trauma pathobiome will elucidate clinical course patterns (recovery and CCI) with microbial composition. The unique biology of the microbiome in different sexes and age groups will require additional subgroup analysis.
Link changes in the microbiome with altered HSPC and erythroid progenitor cells fate establishing gut-bone marrow communication following trauma | 3 years
  We will examine how stress-induced changes following trauma create a pathobiome that modulates HPSC differentiation and maintains altered erythroid progenitor function. The microbiota play a role in both lineage differentiation and also control systemic iron homeostasis by inhibiting intestinal absorption and increasing cellular iron storage. Bone marrow macrophages have a key role in late-stage erythropoiesis by supplying local iron to erythroblasts for hemoglobin production. Isolation of bone marrow macrophages and erythroblasts involved in EBIs and determination of local iron content will define microbiome-induced changes in terminal erythropoiesis.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Mohr, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - UF Academic Research Building, Gainesville, Florida
  - UF Health at Shands Hospital, Gainesville, Florida
  - UF Laboratory of Inflammation Biology and Surgical Science and Shands Hospital at UF, Gainesville, Florida